CLINICAL TRIAL: NCT05611723
Title: Study and Analysis of Biomechanical Parameters of Human Movement Based on Disability Indicators in Older Adults Based on a Multifactorial Analysis: a Cross-sectional Study
Brief Title: Study and Analysis of Biomechanical Parameters of Human Movement Based on Disability Indicators in Older Adults
Acronym: MOBA
Status: Completed | Type: Observational
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: Center for Rehabilitation Research - Polytechnic Institute of Porto (IPP) (Unknown); Universidade do Porto (Other); School of Allied Health Sciences of Porto (ESTSP) - Polytechnic Institute of Porto (IPP) (Other)
Responsible Party: Principal Investigator, Juliana dos Santos Moreira, Master of Science, Polytechnic Institute of Porto
Other Study IDs: CE0064C; 2020.05356.BD (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia, NORTE 2020, FSE EU); UIDB/05210/2020 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia, Portugal and EU)
Record Dates: First submitted 2022-07-06; First posted 2022-11-10 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Disability
Keywords: Aged; Older Adults; Aging; Disability; Disability Evaluation; Biomechanical Phenomena; Biomechanical analysis; Kinematics; Kinetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy older Adults: Healthy older Adults: older adults without disability indicators
- Disability Older Adults: Disability Older Adults: older adults with disability indicators
  Interventions: Other: Exposure to disability

INTERVENTIONS:
Other: Exposure to disability — Disability status assessed by functional measures
  Groups: Disability Older Adults

SUMMARY:
Older adults develop modifications in the execution of movement that lead to impairments in activities of daily living performance. Accordingly, there is a need for technological advances in devices that assist older adults targeting improvements in parameters of movement performance that have the highest impact on the skills of daily living. Therefore, to gather the parameters of movement impacting daily living activities, the main goal of this study is to perform a comparative analysis of the biomechanical movement parameters between older adults with and without disability, performing the tasks: gait, sit-to-stand, timed up and go, quiet standing and climb and descend stairs.

This work was supported by theFundação para a Ciência e Tecnologia (FCT), [grant number 2020.05356.BD] and through R&D Units funding [UIDB/05210/2020], Fundação para a Ciência e Tecnologia (FCT), Portugal and the European Union.

ELIGIBILITY:
Inclusion Criteria:

* older adults, 60 years or over;
* community-dwelling;
* able to perform the tasks (gait, sit-to-stand, climb and descend stairs) independently;

Exclusion Criteria:

* older adults who are institutionalized;
* older adults who have established diagnosis of malignancy or terminal diseases with an anticipated survival of less than 1 year;
* older adults who have stroke history, cerebral hemorrhage, head trauma, or Parkinson's disease;
* older adults who have cognitive impairment, specifically Mini Mental State Examination (Portuguese version) score of 22 for 0 to 2 years of literacy, 24 for 3 to 6 years of literacy and 27 for more than 6 years of literacy (Morgado et al., 2009);
* older adults who have rheumatic pathologies that interfere with the tasks performance;
* older adults who have diabetic foot, lower limb fracture less than 6 weeks, or other related conditions;
* older adults who have unstable cardiovascular disease, liver or renal function failure;
* older adults who have a body mass index greater than or equal to 30 kg/m2;
* older adults who vestibular and/or audition or vision impairments non corrected that influence the performance of tasks;
* older adults who presence of symptoms at the time of evaluation that influences the participant performance of tasks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Portuguese community-dwelling older adults
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Waveforms from full-body joint angles | During tasks performance
  Waveforms from full-body joint angles measured in degrees (°)
Waveform from full-body angular joint velocities | During tasks performance
  Waveform from angular joint velocities measured in degrees per second (°/s)
Waveform from lower limb joint moments | During tasks performance
  Waveform from lower limb joint moments measured in Newton-meter (kgm²/s²)
Waveform from total body energy | During tasks performance
  Waveform from total body energy measured in joules (J)
Waveform from full-body separate segment energy | During tasks performance
  Waveform from body segment energy un joules (J)
Waveform from lower body joint forces | During tasks performance
  Waveform from lower body joint forces measured in Newton (N)
Waveform from lower body joint power | During tasks performance
  Waveform from lower body joint power measured in Watts
Waveform from centre of mass displacement | During tasks performance
  Waveform from centre of mass displacement in m/s
Waveform from centre of pressure displacement | During tasks performance
  Waveform from centre of pressure displacement in m/s

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rehabilitation Research, School of Health, Polytechnic of Porto, Portugal, Porto, Porto District, Portugal